CLINICAL TRIAL: NCT00243009
Title: Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation for the Treatment of Metastatic Renal Cell Carcinoma
Brief Title: Fludarabine and Total-Body Irradiation in Treating Patients Who Are Undergoing a Donor Stem Cell Transplant for Metastatic Kidney Cancer That Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a lack of a referal base, study was terminated.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000447207; OHSU-ONC-03077-L (Other: OHSU Knight Cancer Institute); OHSU-1282 (Other: OHSU IRB)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2010-06

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine, and radiation therapy before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine together with total-body irradiation works in treating patients who are undergoing a donor stem cell transplant for metastatic kidney cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of nonmyeloablative conditioning comprising fludarabine and total-body irradiation followed by allogeneic hematopoietic stem cell transplantation, in terms of 6-month and 12-month response rate, in patients with unresectable metastatic renal cell carcinoma.

OUTLINE:

* Nonmyeloablative conditioning regimen: Patients receive fludarabine IV on days -4 to -2 and total-body irradiation (TBI) on day 0.
* Allogeneic hematopoietic stem cell transplantation (AHSCT): After TBI, patients undergo AHSCT on day 0.
* Immunosuppression: Patients receive oral cyclosporine twice daily on days -3 to 56 followed by a taper until day 81. Patients also receive oral mycophenolate mofetil twice daily on days 0-27 (if patient has a related donor) OR three times daily on days 0-29 and then twice daily on days 30-149 followed by additional tapering until day 180 (if patient has an unrelated donor).

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma, including 1 of the following subtypes:

  * Clear cell
  * Papillary
  * Medullary
* Metastatic disease
* Not amenable to curative surgery
* No CNS metastases

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 6 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* AST or ALT < 4 times ULN

Renal

* Creatinine clearance > 50 mL/min

Cardiovascular

* LVEF > 35%
* No symptomatic congestive heart failure

Pulmonary

* DLCO > 40% of predicted OR
* Total lung capacity or FEV_1 > 30% of predicted

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 30 days since prior biologic therapy

Chemotherapy

* More than 30 days since prior chemotherapy

Radiotherapy

* More than 30 days since prior radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial response) at 6 and 12 months after transplantation

SECONDARY OUTCOMES:
Severity of graft-vs-host-disease by Glucksburg Scale after transplantation for up to 5 years
Incidence of graft rejection based on donor chimerims after transplantation for up to 5 years
Non-relapse mortality as assessed by Kaplan-Meier after transplantation for up to 5 years
Disease-free survival as assessed by Kaplan-Meier after transplantation for up to 5 years
Overall survival as assessed by Kaplan-Meier after transplantation for up to 5 years
Toxicity as measured by CTC AE v 3.0 100 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M. Hayes-Lattin, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States